CLINICAL TRIAL: NCT04162418
Title: A Non-RanDomized Pilot Study of the TEmporary Spur StEnt System for the Treatment of Lesions Located in the InfraPoplitEal ARteries Using a LIMUS-base Drug-coated Balloon (DEEPER LIMUS)
Brief Title: A Study of the TEmporary Spur StEnt System for the Treatment of Lesions Located in the InfraPoplitEal ARteries Using a LIMUS-base DCB
Acronym: DEEPER LIMUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReFlow Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-005
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
Keywords: peripheral arterial disease; critical limb ischemia; infrapopliteal disease
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Treatment with Temporary Spur Stent System and a commercially available, limus-base, drug coated balloon
  Interventions: Device: Temporary Spur Stent System

INTERVENTIONS:
Device: Temporary Spur Stent System — Treatment of qualifying infrapopliteal lesions with Temporary Spur Stent System and a commercially available, limus-base drug-coated balloon

SUMMARY:
This is a non-randomized, prospective, single center pilot study designed to evaluate the safety of the Temporary Spur Stent System to treat patients with infrapopliteal arterial disease, when used in conjunction with a commercially available limus-base drug coated balloon.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide informed consent and able to comply with the study protocol.
2. Life expectancy >1 year in the investigator's opinion.
3. Subject is > 18 years of age.
4. Subjects must have symptoms of limb ischemia, determined by clinical symptoms of Rutherford class 3-5, including severe, life-limiting claudication (R 3), rest pain (R 4), and/or minor tissue loss (R5), that in the opinion of the investigator are not amenable to conservative medical therapy and require endovascular intervention for alleviation of symptoms and tissue preservation
5. Stenotic, restenotic, or occlusive lesions located in the infrapopliteal vessels, with target lesion that can be successfully crossed with a guidewire.
6. Target lesion must meet lesion-specific criteria in pre-screening by angiography at time of procedure (prescreening with CTA, MRA or selective angiography may be performed prior to the index procedure).
7. Target vessel(s) reconstitute(s) at or above the ankle, with the target treated segment extending no more than 10 mm beyond the ankle.

   Note:

   If the anterior tibial or posterior tibial arteries are treated, there must be inline flow to the foot.

   If the peroneal artery is treated, there must be at least one collateral supplying the foot.
8. Target lesion must begin no higher than the tibial trifurcation (popliteal artery excluded).
9. Target vessel reference diameter is measured to be between 2.0 mm to 4.5 mm in diameter, assessed by one of the following methods after successful completion of guidewire crossing of the lesion site:

   1. Intravascular Ultrasound (IVUS)
   2. Optical Coherence Tomography (OCT)
   3. Quantitative Vascular Angiography (QVA)
10. Lesion length must be > 30 mm and < 200 mm.
11. Only one limb may be enrolled per subject. Up to two vessels may be treated per subject; if required, a second modality may be used for treatment in the non-target infrapopliteal vessel. Any treatment of the non-index vessel must be performed prior to the use of the investigative device and only one artery may be treated with the investigative device
12. The treated segment is defined as the total length of artery treated with the investigational device. Target treatment length is <250 mm with a maximum segment of 200 mm separated by 30 mm of healthy tissue between treated lesions.
13. Successful pre-dilatation of the target lesion as outlined in the procedure instructions, defined as resulting in stenosis <50%, without resulting flow limiting (Type D or greater) dissection, thrombus, or aneurysm by angiography prior to the insertion of the investigative device.
14. Iliac, SFA and popliteal inflow lesions can be treated using standard angioplasty and/or drug coated balloon and/or an approved stent (no atherectomy) during the index procedure or >30 days prior. Inflow lesions treated intraprocedure must be treated first, prior to consideration of treatment of infrapopliteal lesions. If pre-screening with duplex ultrasound, angiography, CTA, or MRA has been performed < 365 days prior to the procedure, intra-procedure angiography of the aorto-iliac vasculature is not required, however, the femoropopliteal inflow must still be imaged using angiography during the index procedure. Inflow lesions must have a healthy vessel segment of >30 mm between the study lesion and the treated segment, defined as less than 50% stenosis without aneurysmal segments.
15. Retrograde access (in the infrapopliteal arteries) is permitted for lesion crossing, however, the Temporary Spur Stent System must be deployed from antegrade access.
16. For subjects with bilateral disease, planned treatment of the contralateral limb must either be performed >30 days prior to the index procedure or > 14 days following the index procedure.

Exclusion Criteria:

1. Subject unwilling or unlikely to comply with the appropriate follow up time for the duration of the study in the opinion of the investigator.
2. Subject is pregnant or planning to become pregnant during the course of the trial.
3. Subject has an active infection that is not controlled at the time of the procedure, including septicemia or bacteremia.
4. Subject has osteomyelitis proximal to the phalanges. Osteomyelitis in the digit(s) of the target foot is permitted.
5. Subject has a heel wound, unless osteomyelitis has been ruled out with MRI, MRA, or nuclear medicine bone scan
6. Planned major (above the ankle) amputation of the target limb. A planned or previous minor (transmetatarsal amputation or digit amputation) is permitted
7. Recent myocardial infarction or stroke < 90 days prior to the index procedure.
8. Symptomatic acute heart failure NYHA class III or greater.
9. Impaired renal function (eGFR <25 mL/min) within 30 days of procedure or end stage renal disease on dialysis
10. Subject with vasculitis, systemic Lupus Erythematosus or Polymyalgia Rheumatica.
11. Subject receiving chronic or intravenous corticosteroid therapy.
12. Inability to tolerate dual antiplatelet and/or anticoagulation therapy.
13. Known allergies or sensitivities to heparin, antiplatelet drugs, other anticoagulant therapies which could not be substituted, drug balloon coatings and their excipients, including, but not limited to, paclitaxel, sirolimus, or zotarolimus, or an allergy to contrast media that cannot be adequately pre-treated prior to the index procedure.
14. The subject is currently enrolled in another investigational device or drug trial that interferes with the study endpoints.
15. Known allergy to nitinol or nickel.
16. Prior stent(s) within the target vessel, or bypass surgery of or within the target vessel(s)
17. Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion. Inflow must also be free of aneurysmal segments.
18. Previous treatment failure of inflow arteries (Iliac, SFA and popliteal) which required a surgical procedure. Prior bypass above the level of the infrapopliteal arteries is permitted.
19. Previous treatment of inflow lesions, if not treated during the index procedure, must have been performed >30 days prior to the index procedure.
20. Previous treatment of the target vessel <30 days prior to index procedure
21. Angiographic evidence of thrombus within target limb.
22. Inability to obtain antegrade access in the limb from which the investigative device can be deployed.
23. Extremely severe calcification classified as grade 4 as measured by the Peripheral Academic Research Consortium (PARC) score or the Peripheral Arterial Calcium Scoring System (PACSS) that, in the investigator's opinion, would not be amenable to PTA (see Appendix I for definitions).
24. Type D dissections or greater incurred during predilation or CTO crossing (see Appendix I for definitions).
25. Significant (>50%) stenosis of inflow arteries or unsuccessful treatment of inflow lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of All-Cause Mortality, Major Amputation and Clinically Driven Target Lesion Revascularization (CD-TLR) at 6 months | 6 months
  6 month composite of All-Cause Mortality, Major Amputation and Clinically Driven Target Lesion Revascularization (CD-TLR)

SECONDARY OUTCOMES:
Secondary Efficacy: Late lumen loss | 6 months
  Late Lumen Loss (LLL) of the target lesion by angiogram/QVA at 6 months
Secondary Efficacy: Primary Patency | 6 months
  2. Primary patency (flow/no flow) of treated lesion sites by angiogram/QVA in subjects who are free from CD-TLR at 6 months.
Secondary Efficacy: Rutherford class | 12 months
  The second secondary efficacy measurement is change in Rutherford class score at 3, 6 and 12 months. Rutherford score is a classification system for patients with peripheral vascular disease.
  Categories are numbered from 0 to 6, with 0 being asymptomatic, and 6 being major tissue loss, functional foot no longer salvageable. Higher values are therefore considered a worse outcome.
  Rutherford class zero: No symptoms; Rutherford class 1: Mild Claudication (minimal leg pain with ambulation) symptoms; Rutherford Class 2: Moderate Claudication (moderate leg pain with ambulation); Rutherford Class 3: Severe claudication (severe leg pain with ambulation); Rutherford Class 4: Ischemic Rest pain (leg pain at rest); Rutherford Class 5: Minor tissue loss (nonhealing ulcer, focal gangrene, diffuse pedal ischemia); Rutherford class 6: Major tissue loss (extending above the transmetatarsal TM level, functional foot no longer salvageable.
Secpndary Efficacy: Wound healing | 12 months
  The third secondary efficacy endpoint is wound healing for subjects with Rutherford class 5 at 6 and 12 months, as assessed by the investigator using WIfI score and descriptive characteristics, including change in wound size measured by any decrease in wound surface area.
  The WIfI classification scoring system is a grading system using a composite score of wound (W), ischemia (I), and foot infection (fi). These three different categories are graded from 0 to 3 with 0 being the best and 3 being the worst.
  The total score will be provided (clinical stage 1-5), which is used to estimate the risk for major amputation at one year. Patients with a score of 1 are considered low risk, and patients with a score of 5 are considered high risk (foot not salvageable). Therefore, higher values are considered a worse outcome.
  The composite score is calculated by adding up the score from each category.

OTHER OUTCOMES:
Secondary Safety: 30 days | 30 days
  1. Freedom from target limb Major Adverse Limb Event (MALE) & All- cause perioperative death (POD) at 30 days
Secondary Safety: 6 and 12 months | 12 months
  Freedom from MALE of the target limb at 6 and 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — Univ-Klinikum LKH Graz
Locations (1):
- Univ.-Klinikum LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
No plan for sharing of IPD